CLINICAL TRIAL: NCT01650753
Title: Quantitative Evaluation of the Colonization and Persistence of Bifidobacterium Longum Ssp Longum AH1206 in the Gastrointestinal Tract and Its Tolerance by Human Subjects
Brief Title: Colonization and Persistence of Bifidobacterium Longum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Responsible Party: Principal Investigator, Jens Walter, PhD: Department of Food Science and Technology, University of Nebraska Lincoln
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UNL 222-12 FB
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Bacterium; Agent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic Powder (Experimental): Probiotic: Bifidobacterium longum subsp longum AH1206
  Interventions: Dietary Supplement: Probiotic Powder
- Placebo Powder (Placebo Comparator): Equivalent amount (same volume) of maltodextrin
  Interventions: Dietary Supplement: Placebo powder

INTERVENTIONS:
Dietary Supplement: Probiotic Powder — Bifidobacterium longum subsp longum AH1206 freeze dried and provided as a powder in a sachet (10^10 cells/sachet)
  Arms: Probiotic Powder
Dietary Supplement: Placebo powder — powdered maltodextrin inthe same volume and the freeze dried probiotic in a similar size sachet
  Arms: Placebo Powder

SUMMARY:
Healthy adults referred to as the absence of intestinal disorders, liver and kidney problems, lactose intolerance, and no use of ongoing medication for chronic diseases will be recruited. This research study will test the persistence of the probiotic (healthy bacterial) strain Bifidobacterium longum spp. longum in the human gastrointestinal tract after it is consumed, how it is tolerated, and its interactions with other micro-organisms already present in your gastrointestinal tract. The strain used is similar to bacteria used in probiotic yogurts, and the species Bifidobacterium is generally regarded as safe. The patient will be asked to will be consume a probiotic powder containing Bifidobacterium longum spp. longum strain AH1206 and a placebo in a random order, with neither the patient nor the investigators knowing the identity of the preparations given. Persistence or presence of the probiotic strain will be based on analysis of fecal (stool or bowel movement) samples provided.

DETAILED DESCRIPTION:
The study will be performed as a 14 week randomized crossover trial with two treatments, one of which is the placebo. The randomization design will be provided by collaborators at Mead Johnson, and the study will be performed double blinded, such that no study staff will be informed about the nature of the product. Each treatment period will consist of a one week baseline period, in which one fecal sample will be collected. This will be followed by a two week feeding period in which the probiotic will be administered at a constant dose of 10^10 cells per day in 50 to 100 ml of either cold or room temperature tab water. At day 7 and 14 (last day of feeding), a fecal sample will be collected. The last sample during feeding will also serve as day 0 of Test of Persistence (TOP) period. Persistence of the probiotic strains will be tested during the TOP period at day 4, 8, 16, and 28 (4 weeks) for a total of 7 fecal samples. The subjects will then crossover to the other treatment and the above fecal sample collections will be repeated. Fecal samples will be provided by the subjects using disposable stool collection containers not longer than 2 hours after defecation. In the lab fecal samples will be stored undiluted (four aliquots) and as 1/10 dilutions in PBS buffer (four aliquots). The investigators will also prepare five tubes with 1 gram aliquots of each fecal sample and will provide these samples de-identified to Mead Johnson Nutrition for future analyses. Experimental design. Fecal samples will be studied by qRT-PCR. Fecal samples may be subjected to pyrosequencing and selective culturing.

All subjects will fill out a Gastrointestinal Symptom Rating Scale (GSRS) questionnaire (at week GSRS at week 1, 2, 3, 4 and 8, 9, 10 11) to test the acceptance and safety of the strain, and to test if subjects remain eligible for the study. Weeks 1 and 8 are the baseline visits, weeks 4 and 11 are one week after subject stops taking study product. Subjects that have begun or expect to begin antibiotic treatment or that have experienced unacceptable side effects will stop their participation.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent and willingness to participate in the study and comply with its procedures.
* Male or Female
* Aged 19 years of age and over.
* Be in generally good health as determined by the investigators. BMI of 18.5-29.9 kg/m2
* Free of any gastrointestinal disorders or complaints, as determined by the Bowel Disease Questionnaire (Talley et al., 1990), at visit 1.
* Not pregnant and not lactating.
* Be able to provide fecal samples for the duration of the 14 week study.
* Be willing to complete the Gastrointestinal Symptom Rating Scale (GSRS) once a week.

Exclusion Criteria:

* Less than 19 years of age.
* Underweighted or obese based on BMI.
* Antibiotic usage 3 months prior to study or during study.
* Significant acute or chronic existing illness [cardiovascular, gastrointestinal, immunological] or a condition which in the investigators judgment, contraindicates involvement in the study.
* Prior gastrointestinal surgery (apart from appendicectomy and hernia repair) or recent unexplained bleeding which, in the Investigator's judgment, contraindicates participation in the study.
* Having a condition or taking a medication, dietary supplement or food product (e.g. probiotic yogurt) that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results.
* Individuals who, in the opinion of the investigator, are considered to be poor clinical attendees or unlikely for any reason to be able to comply with the trial.
* Patients receiving treatment involving experimental drugs.
* Pregnant or lactating.
* Participation in a recent experimental trial less than 30 days prior to this study.
* Have a malignant disease or any concomitant end-stage organ disease, which, in the Investigator's judgment, contraindicates participation in the study.
* Inability to provide fecal samples for the duration of the 14 week study.
* Inability to complete the weekly GSRS.se on antibiotics, suppressed immune systems

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Persistence or presence of the probiotic strain Bifidobacterium Longum ssp longum AH1206. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jens Walter, PhD, Principal Investigator — University of Nebraska Lincoln